CLINICAL TRIAL: NCT01163747
Title: A Randomized, Parallel-group, Open-label, Multicenter Study to Evaluate the Effects of Tocilizumab on Vaccination in Subjects With Active Rheumatoid Arthritis Receiving Background Methotrexate
Brief Title: A Study of the Effects of RoActemra/Actemra on Vaccination in Patients With Rheumatoid Arthritis on Background Methotrexate (VISARA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA25256
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Results first posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate; 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines

ARMS (2):
- Methotrexate (Active Comparator): Participants continued to receive their standard dose of methotrexate up to Week 8. From Week 8 participants also received 8 mg/kg tocilizumab intravenously every 4 weeks until Week 20. At Week 3 participants received both pneumococcal and tetanus toxoid vaccinations.
  Interventions: Biological: tocilizumab; Drug: methotrexate; Biological: 23-Valent Pneumococcal Polysaccharide Vaccine; Biological: Tetanus Toxoid Adsorbed Vaccine
- Tocilizumab + Methotrexate (Experimental): Participants received 8 mg/kg tocilizumab intravenously at Baseline (Day 1) and every 4 weeks up to Week 20, in addition to their standard dose of methotrexate. At Week 3 participants received both pneumococcal and tetanus toxoid vaccinations.
  Interventions: Biological: tocilizumab; Drug: methotrexate; Biological: 23-Valent Pneumococcal Polysaccharide Vaccine; Biological: Tetanus Toxoid Adsorbed Vaccine

INTERVENTIONS:
Biological: tocilizumab — Intravenous repeating dose
  Other Names: RoActemra; Actemra
Drug: methotrexate — A stable dose of between 7.5 and 25 mg/week, oral or parenteral.
Biological: 23-Valent Pneumococcal Polysaccharide Vaccine — Intramuscular or subcutaneous injection
  Other Names: Pneumovax
Biological: Tetanus Toxoid Adsorbed Vaccine — Intramuscular injection

SUMMARY:
This randomized, parallel-group, open-label study will evaluate the effect of Actemra (tocilizumab) on vaccination in patients with active rheumatoid arthritis who have an inadequate response to methotrexate and who have had an inadequate clinical response or were intolerant to treatment with one or more anti-tumor necrosis factor (anti-TNF) therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 to < 65 years of age
* Rheumatoid Arthritis (RA) of > 6 months duration at baseline (American College of Rheumatology criteria)
* Willing to receive immunization with pneumococcal polysaccharide and tetanus toxoid adsorbed vaccines
* Previous immunization with pneumococcal polysaccharide must have occurred ≥ 3 years of baseline, with tetanus containing vaccine ≥ 5 years
* Methotrexate therapy for at least 8 weeks prior to baseline at stable dose of 7.5-25 mg/week (oral or parenteral)
* Other disease-modifying antirheumatic drugs (DMARDs) must be withdrawn before baseline
* Oral corticosteroids must be at stable dose of < 10 mg/day prednisone or equivalent
* Body weight ≤ 150 kg at screening

Exclusion Criteria:

* Major surgery (including joint surgery) within 12 weeks prior to baseline or planned major surgery within 8 weeks after baseline
* History of or current inflammatory joint disease or rheumatic autoimmune disease other than RA
* Pre-existing central nervous system demyelinating or seizure disorders
* Active current or history of recurrent bacterial, viral fungal, mycobacterial and other infections
* Any major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks prior to baseline or oral antibiotics within 2 weeks prior to baseline
* Active tuberculosis requiring treatment within 3 years prior to baseline
* Primary or secondary immunodeficiency (history or currently active)
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* Previous treatment with RoActemra/Actemra

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micki Klearman, M.D., Study Director — Genentech, Inc.
Locations (45):
- United States (45):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Fullerton, California
  - Hemet, California
  - San Leandro, California
  - Santa Maria, California
  - Upland, California
  - Bridgeport, Connecticut
  - Melbourne, Florida
  - South Miami, Florida
  - Tavares, Florida
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Maywood, Illinois
  - Vernon Hills, Illinois
  - South Bend, Indiana
  - Baltimore, Maryland
  - Saint Clair Shores, Michigan
  - Tupelo, Mississippi
  - Las Vegas, Nevada
  - Manalapan, New Jersey
  - Albany, New York
  - Belmont, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Cleveland, Ohio
  - Gallipolis, Ohio
  - Middleburg Heights, Ohio
  - Lake Oswego, Oregon
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wexford, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Orangeburg, South Carolina
  - Dallas, Texas
  - Mesquite, Texas
  - Tacoma, Washington
  - Clarksburg, West Virginia

REFERENCES:
- [Result] Bingham CO 3rd, Rizzo W, Kivitz A, Hassanali A, Upmanyu R, Klearman M. Humoral immune response to vaccines in patients with rheumatoid arthritis treated with tocilizumab: results of a randomised controlled trial (VISARA). Ann Rheum Dis. 2015 May;74(5):818-22. doi: 10.1136/annrheumdis-2013-204427. Epub 2014 Jan 21. PMID 24448345

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 35 centers in the United States. Among the 112 patients screened, 91 patients were randomized in a 1:2 ratio to the methotrexate alone or to the tocilizumab + methotrexate treatment group.
Period: Overall Study
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Started | 31 | 60
Per Protocol Population | 27 (Participants who received at least 1 dose of study treatment excluding major protocol violators.) | 54 (Participants who received at least 1 dose of study treatment excluding major protocol violators.)
Completed | 25 | 49
Not Completed | 6 | 11
Not completed — Adverse Event | 0 | 5
Not completed — Insufficient Therapeutic Response | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Refused Treatment | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Tocilizumab + Methotrexate | Total
Number analyzed (Participants) | 27 | 54 | 81
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the per protocol population.
  years | 51.4 (9.47) | 51.1 (8.90) | 51.2 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 41 | 63
  Male | 5 | 13 | 18
Region of Enrollment [Number; unit: participants]
  United States | 27 | 54 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Responded to ≥ 6 of 12 Anti-pneumococcal Antibody Serotypes
Description: Serum levels of antibody to pneumococcal vaccine were drawn 5 weeks after vaccination with 23-valent pneumococcal polysaccharide vaccine to assess humoral immune response. A positive response to the pneumococcal vaccine was defined as a 2-fold increase in serum antibody titers from Baseline or an increase of > 1 mg/L from Baseline levels.
  The 12 serotypes evaluated were pneumococcal serotypes 1, 3, 4, 6B, 8, 9N, 12F, 14, 19F, 23F, 7F, and 18C.
Time Frame: Baseline (Week 3) and Week 8 (5 weeks post-vaccination)
Population: Evaluable per protocol population for pneumococcal polysaccharide vaccine: participants who received at least one dose of study medication, had no major protocol violations, had both baseline (Week 3) and Week 8 assessments of response with evaluable titers to the pneumococcal vaccine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 24 | 50
percentage of participants | 70.8 [52.6 to 89.0] | 60.0 [46.4 to 73.6]

2. Secondary Outcome: Percentage of Participants Who Responded to Combinations of 12 Anti-Pneumococcal Antibody Serotypes
Description: as for outcome 1
Time Frame: Baseline (Week 3) and Week 8 (5 weeks post-vaccination)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 24 | 50
percentage of participants
  Responded to ≥1 out of 12 serotypes | 87.5 [74.3 to 100.0] | 90.0 [81.7 to 98.3]
  Responded to ≥2 out of 12 serotypes | 87.5 [74.3 to 100.0] | 86.0 [76.4 to 95.6]
  Responded to ≥3 out of 12 serotypes | 83.3 [68.4 to 98.2] | 80.0 [68.9 to 91.1]
  Responded to ≥4 out of 12 serotypes | 83.3 [68.4 to 98.2] | 74.0 [61.8 to 86.2]
  Responded to ≥5 out of 12 serotypes | 83.3 [68.4 to 98.2] | 66.0 [52.9 to 79.1]
  Responded to ≥6 out of 12 serotypes | 70.8 [52.6 to 89.0] | 60.0 [46.4 to 73.6]
  Responded to ≥7 out of 12 serotypes | 58.3 [38.6 to 78.1] | 54.0 [40.2 to 67.8]
  Responded to ≥8 out of 12 serotypes | 58.3 [38.6 to 78.1] | 38.0 [24.5 to 51.5]
  Responded to ≥9 out of 12 serotypes | 45.8 [25.9 to 65.8] | 32.0 [19.1 to 44.9]
  Responded to ≥10 out of 12 serotypes | 29.2 [11.0 to 47.4] | 20.0 [8.9 to 31.1]
  Responded to ≥ 11 out of 12 serotypes | 20.8 [4.6 to 37.1] | 12.0 [3.0 to 21.0]
  Responded to 12 out of 12 serotypes | 8.3 [0.0 to 19.4] | 6.0 [0.0 to 12.6]

3. Secondary Outcome: Percentage of Participants With a Positive Response to Tetanus Toxoid Vaccination
Description: A positive response to the tetanus toxoid vaccination was defined as antibody levels ≥ 0.2 IU/mL for participants with Baseline tetanus antibody levels < 0.1 IU/mL, or a 4-fold increase in antibody levels compared with Baseline for participants with Baseline tetanus antibody levels ≥ 0.1 IU/mL.
Time Frame: Baseline (Week 3) and Week 8 (5 weeks post-vaccination)
Population: Evaluable per protocol population for tetanus toxoid vaccine: participants who received at least one dose of study medication, had no major protocol violations, had both baseline (Week 3) and Week 8 assessments of response with evaluable titers to the tetanus toxoid vaccine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 23 | 50
percentage of participants | 39.1 [19.2 to 59.1] | 42.0 [28.3 to 55.7]

4. Secondary Outcome: Change From Baseline in Levels of Anti-pneumococcal Antibody 5 Weeks After Vaccination
Description: Levels of anti-pneumococcal antibodies were measured by a central laboratory from serum samples taken prior to vaccination (Week 3) and 5 weeks post vaccination (Week 8).
Time Frame: Baseline (Week 3) and Week 8 (5 weeks post-vaccination)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 22 | 48
mg/L
  Baseline | 91.1 (122.91) | 73.9 (63.50)
  Week 8 | 307.2 (270.25) | 184.2 (197.99)
  Change from Baseline | 216.1 (261.85) | 110.2 (188.74)

5. Secondary Outcome: Change From Baseline in Levels of Anti-tetanus Antibody 5 Weeks After Vaccination
Description: Levels of anti-tetanus antibodies were measured by a central laboratory from serum samples taken prior to vaccination (Week 3) and 5 weeks post vaccination (Week 8).
Time Frame: Baseline (Week 3) and Week 8 (5 weeks post-vaccination)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 23 | 50
IU/mL
  Baseline | 2 (1.3) | 2 (1.9)
  Week 8 | 9 (12.4) | 9 (9.2)
  Change from Baseline | 7 (12.3) | 7 (9.0)

6. Secondary Outcome: Percentage of Participants Who Responded to Each of the 12 Anti-Pneumococcal Antibody Serotypes
Description: Serum levels of antibody to pneumococcal vaccine were drawn 5 weeks after vaccination with 23-valent pneumococcal polysaccharide vaccine to assess humoral immune response. A positive response to the pneumococcal vaccine was defined as a 2-fold increase in serum antibody titers from Baseline or an increase of > 1 mg/L from Baseline levels.
  The 12 serotypes evaluated were pneumococcal serotypes 1, 3, 4, 6B, 7F, 8, 9N, 12F, 14, 18C, 19F and 23F.
Time Frame: Baseline (Week 3) and Week 8 (5 weeks post-vaccination)
Population: Evaluable per protocol population for pneumococcal polysaccharide vaccine. N indicates the number of participants with available data for each serotype. No imputation was performed.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 24 | 50
percentage of participants
  Serotype 1 response [N=24, 49] | 79.2 | 65.3
  Serotype 3 response [N=24, 49] | 62.5 | 53.1
  Serotype 4 response [N=24, 50] | 33.3 | 38.0
  Serotype 6B response [N=24, 50] | 58.3 | 46.0
  Serotype 7F response [N=24, 49] | 66.7 | 61.2
  Serotype 8 response [N=24, 49] | 75.0 | 59.2
  Serotype 9N response [N=23, 50] | 73.9 | 56.0
  Serotype 12F response [N=23, 49] | 21.7 | 26.5
  Serotype 14 response [N=21, 50] | 57.1 | 56.0
  Serotype 18C response [N=24, 50] | 79.2 | 64.0
  Serotype 19F response [N=24, 50] | 70.8 | 54.0
  Serotype 23F response [N=24, 50] | 50.0 | 44.0

7. Secondary Outcome: Number of Participants With Adverse Events Through Week 8
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A Serious Adverse Event (SAE) is any AE that is fatal or is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: 8 weeks
Population: All participants who received at least one dose of study treatment were included in the safety evaluation.
Measure: Number; unit: participants
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 31 | 60
participants
  Any adverse event | 3 | 23
  Serious adverse event | 1 | 2
  Deaths | 0 | 0
  Withdrawals due to adverse events | 0 | 1

ADVERSE EVENTS:
Time Frame: From Day 1 through Week 28.
Arm/Group | Methotrexate | Tocilizumab + Methotrexate
Serious Adverse Events (participants affected / at risk) | 1/31 | 3/60
Other Adverse Events (participants affected / at risk) | 9/31 | 25/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=31) | Tocilizumab + Methotrexate (N=60)
Cellulitis (Infections and infestations) | 1 | 1
Intraspinal abscess (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=31) | Tocilizumab + Methotrexate (N=60)
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Sinusitis (Infections and infestations) | 1 | 5
Nasopharyngitis (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.